CLINICAL TRIAL: NCT06410573
Title: The Effect Of Self-Breast Examination Training Provided To Women Between 18 And 49 Years Of Age And Practice On The Belief Of Breast Health: A Randomized Controlled Study
Brief Title: The Effect Of Self-Breast Examination Training On The Belief Of Breast Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KaratayUH9
Record Dates: First submitted 2023-06-01; First posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Women of Reproductive Age
Keywords: Neoplasms; Early Detection of Cancer; Breast Neoplasms; health education
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Health Education

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training on Breast Self-Examination (Experimental): In the training, women will be divided into 5 groups and the training will be held in 5 separate sessions in one day. A training program will be completed with 9 women. All trainings will be conducted under the same conditions in the school's training room. Before the training, women will be informed about the training and their permission and consent will be obtained. The training prepared by the researcher will be presented to the women in the experimental group of the study. The presentation used in the training will include information about breast cancer, breast cancer screening programs and breast self-examination.
  Interventions: Behavioral: Breast Self-Examination and Practice
- Control (No Intervention): 1 week follow-up.

INTERVENTIONS:
Behavioral: Breast Self-Examination and Practice — In the training, women will be divided into 5 groups and the training will be held in 5 separate sessions in one day. A training program will be completed with 9 women. All trainings will be conducted under the same conditions in the school's training room. Before the training, women will be informed about the training and their permission and consent will be obtained. The training prepared by the researcher will be presented to the women in the experimental group of the study. The presentation used in the training will include information about breast cancer, breast cancer screening programs and breast self-examination. In the presentation, the steps of breast self-examination will be shown step by step using visual materials.
  Arms: Training on Breast Self-Examination

SUMMARY:
The aim of the present research was to detect the effect of self-breast examination provided to women between 18 and 49 years of age and practice on the belief of women on their breast health.

DETAILED DESCRIPTION:
The aim of this study was to investigate the effect of breast self-examination training and practice on breast health beliefs. The study was a pretest-posttest randomized controlled experimental design. Women in the experimental group of the study will be provided with the training prepared by the researcher. The presentation used in the training will include information about breast cancer, breast cancer screening programs and breast self-examination. In the presentation, the steps of breast self-examination were shown step by step using visual materials. In addition to the slide presentation about breast cancer and breast self-examination, women will be trained on breast self-examination with a breast examination model using the "show first, then do it" training technique, and the accuracy will be confirmed by asking women to do it. By using the model in breast examination, it will be determined what women do right and what they do wrong during the examination. Data will be collected with Personal Information Form and Champion Health Belief Model Scale.

ELIGIBILITY:
Inclusion Criteria:

* Fertility process to continue
* No communication problems
* Not having a disease that will affect perception

Exclusion Criteria:

* Having been previously diagnosed with breast cancer or receiving breast cancer treatment
* Being diagnosed with a medical mental illness and receiving treatment for this reason
* Being under active treatment in hospital due to any problem

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2022-11-06 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Breast Self-Examination Training and Breast Health Beliefs | 1 month will be followed
  This outcome is assessed with the Champion Health Belief Model Scale. A higher score on the scale indicates an increase in sensitivity and caring, a higher perception of benefits for the perception of benefits, and a higher perception of obstacles for the perception of obstacles.

CONTACTS AND LOCATIONS:
Locations (1):
- KTO Karatay University, Konya, Karatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided